CLINICAL TRIAL: NCT05149924
Title: A Multicenter, Randomized, Single-blind, Active-controlled, Phase III Clinical Study to Compare the Efficacy and Safety of QL1012(Recombinant Human Follicle-stimulating Hormone) and Gonal-f ® in Women Undergoing Controlled Ovarian Hyperstimulation for Assisted Reproductive Treatment
Brief Title: Efficacy and Safety of QL1012 in Women for Assisted Reproductive Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QL1012-002
Record Dates: First submitted 2021-11-12; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1012，Recombinant Human Follicle Stimulating Hormone for Injection (Experimental)
  Interventions: Drug: QL1012
- Gonal-f ® (Active Comparator)
  Interventions: Drug: Gonal-f ®

INTERVENTIONS:
Drug: QL1012 — Subcutaneous injection,starting dose within 75IU ~ 300IU determined by the age , maximum daily dose 450IU
  Arms: QL1012，Recombinant Human Follicle Stimulating Hormone for Injection
Drug: Gonal-f ® — Subcutaneous injection,starting dose within 75IU ~ 300IU determined by the age , maximum daily dose 450IU
  Arms: Gonal-f ®

SUMMARY:
The study is conducted to confirm equivalence between QL1012 (a new biosimilar formulation of Recombinant Human Follicle-stimulating Hormone) and Gonal-f® with respect to the number of oocytes retrieved in women for assisted reproductive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Aged 20 ~ 39 years(inclusive)
3. Body mass index (BMI) between 18~30 kg/m2(inclusive)
4. Regular menstrual cycle (25~35 days)
5. Basal FSH < 10 IU/L (menstrual cycle day 2~5)

Exclusion Criteria:

1. History of ≥3 previously completed IVF/ICSI-ET cycles without clinical pregnancy
2. History of ≥3 recurrent spontaneous miscarriages
3. Patients with high risk of ovarian hyperstimulation syndrome (OHSS)
4. Primary ovarian failure or poor responders to ovarian stimulation
5. Presence of pregnancy in previous 3 months
6. Presence of clinically significant systemic disease, endocrine disease or metabolic abnormalities
7. History of malignant tumors of the ovary, breast, uterus, hypothalamus, pituitary gland, etc.;

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 36-38 hours after hCG administration
  36-38 hours after hCG administration, transvaginal ultrasound-guided aspiration was performed as required, and the number of oocytes was recorded.

SECONDARY OUTCOMES:
Total dose of r-hFSH administered | From date of randomization up to 16 days
Number of days of r-hFSH stimulation | From date of randomization up to 16 days
Serum estradiol concentration | From date of randomization up to 16 days
Endometrial thickness | From date of randomization up to 16 days
Fertilization Rate of Oocytes | Day 1 of IVF/ICSI
Rate of high-quality embryos | 3 days after oocyte retrieval
Implantation rate | five to six weeks after oocyte retrieval
clinical pregnancy rate | 35 ± 4 days after embryo transfer
Ongoing pregnancy rate | Ten weeks after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China